CLINICAL TRIAL: NCT05973188
Title: Safety and Efficacy of Rivaroxaban and Apixaban in Comparison to Warfarin in Left Ventricular Clot- a Clinical Trial
Brief Title: Safety and Efficacy of Rivaroxaban and Apixaban in Comparison to Warfarin in Left Ventricular Clot- Clinical Trial
Acronym: WRAP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peshawar Institute of Cardiology (Other Government)
Collaborators: Getz Pharma (Industry)
Responsible Party: Principal Investigator, Dr. Ihsan Ullah, Doctor, Peshawar Institute of Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRC/23/09
Record Dates: First submitted 2023-05-08; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Left Ventricular Thrombus
Keywords: Left ventricular thrombus, warfarin, rivaroxaban, apixaban
MeSH Terms: interventions — Warfarin; Rivaroxaban; apixaban; Tablets

STUDY DESIGN:
Intervention Model Description: Randomized and open label. We will randomly assign first patient into group A that is control group (warfarin group) then next patient to group B (rivaroxaban group) and then next patient into group C (Apixaban group). We will repeat the cycle to achieve the target sample size in each group. Patients will be randomized in group A, B and C in a ratio of 1:1:1, to either control group A (Warfarin group with dose adjusted, target INR 2-3), group B (Rivaroxaban 20mg QD) and group C (Apixaban 5mg BD or 2.5mg BD if having two or more of the following, patients with age ≥80years and/or creatinin≥1.5 and/or body weight ≤60kg). LVT resolution will be assessed by blinded cardiologist via transthoracic echocardiogram at 1, 3 and 6 months' interval after starting on the respective regimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A, warfarin group (Active Comparator): Patients started on warfarin, dose will be adjusted according to patient target INR (2-3)
  Interventions: Drug: Warfarin
- Group B, Rivaroxaban (Xcept) (Experimental): Patients started on rivaroxaban 20mg single dose in 24hours
  Interventions: Drug: Rivaroxaban 20 MG Oral Tablet
- Group C, Apixaban ( Apixaget) (Experimental): Patients started on Apixaban 5mg or 2.5mg (12hours apart)
  Interventions: Drug: Apixaban 5mg or 2.5mg oral tablet

INTERVENTIONS:
Drug: Warfarin — Anticoagulant
  Other Names: Warfarin oral tablet
  Arms: Group A, warfarin group
Drug: Rivaroxaban 20 MG Oral Tablet — Anticoagulant
  Other Names: Xcept
  Arms: Group B, Rivaroxaban (Xcept)
Drug: Apixaban 5mg or 2.5mg oral tablet — Anticoagulant
  Other Names: Apixaget
  Arms: Group C, Apixaban ( Apixaget)

SUMMARY:
The investigators aimed to design this randomized control trial to compare rivaroxaban and apixaban with warfarin in Left ventricular thrombus resolution by

* Success rate of left ventricular thrombus resolution on follow up echocardiograms to be done at 1st, 3rd and 6th months after starting on these drugs.
* Compare the adverse events of each drug in terms of major bleeding and stroke on follow up.

Left ventricular thrombus (LVT) leads to thromboembolism in about 10-15% cases. Currently, guidelines recommended therapy for LVT is warfarin but treating LVT with warfarin is challenging due to

* Its narrow therapeutic window.
* Drug-drug and drug-food interaction.
* Frequently tested International normalization ratio (INR) and cost effectiveness especially in low to middle income countries.

In contrast Rivaroxaban and Apixaban has no drug-food or major drug-drug interaction and moreover it doesn't require frequent checks on INR and that's the reason Rivaroxaban and apixaban use in LVT is gaining traction over time but there is paucity of data both nationally and internationally. So further studies are required to evaluate the efficacy and safety of rivaroxaban and apixaban in comparison to warfarin in LVT, especially in low to middle income countries.

DETAILED DESCRIPTION:
1. TITLE:

   Safety and efficacy of Rivaroxaban and Apixaban in comparison to Warfarin in Left ventricular clot- clinical trial
2. INTRODUCTION:

   Left ventricular thrombus (LVT) is a known life threatening complication of myocardial systolic dysfunction leading to thromboembolism in about 10-15% cases1. The incidence of LVT has significantly decreased from 40% in pre-reperfusion era to 4% in reperfusion era but still it's a significant number to treat and minimize mortality and morbidities2.3. Up-to-date, guidelines recommended therapy for LVT is warfarin but due to its narrow therapeutic window, drug-drug and drug-food interaction, its use is challenging and cost effective, especially in low to middle income countries as it requires frequent checks on INR (International normalization ratio). In contrast Rivaroxaban has no drug-food or major drug-drug interaction and moreover it doesn't require frequent checks on INR and that's the reason Rivaroxaban use in LVT is gaining traction over time but there is paucity of data both nationally and internationally. Abdelnabi M et al. published the first RCT (randomized control trial, No-LVT trial) on Egyptian population and concluded that rivaroxaban is non inferior to warfarin in LVT but their sample was n=79 out of which rivaroxaban arm had 39 patients only with a power of 80%. Alcalai R et al,4 studied and compared warfarin and Apixaban in LV-thrombus and concluded that Apixaban is non inferior to warfarin in LV-thrombus but their sample size was very low to 17 patients in warfarin and 18 patients in apixaban group. So further studies are required to evaluate the safety and efficacy of rivaroxaban and apixaban in LVT specially in low to middle income countries where LVT management with warfarin is challenging because of narrowed therapeutic window and frequently testing INR. The investigators aimed to design this RCT to compare rivaroxaban and apixaban with warfarin in LVT in terms of safety and efficacy.
3. HYPOTHESIS:

Direct acting oral anticoagulation (rivaroxaban and apixaban) is non inferior to warfarin in LV thrombus resolution

4. MATERIALS AND METHODS: 4a. Study Design: It will be a prospective, randomized, open-label, parallel-group, noninferiority trial to evaluate the efficacy and safety of rivaroxaban and apixaban versus warfarin in the treatment of LVT.

4b. Study Settings: Peshawar Institute of Cardiology (PIC). 4c. Study Duration:

1 year

4d. Sample Size:

Type: Binary Yes/No Type Variable (e.g. response vs no response) Design: Parallel Group Objective: Non-inferiority

* Group 1 (Warfarin group): 48%
* Group 2 (Rivaroxaban group): 72%
* Group 3 (Apixaban group):

Non-inferiority criteria: 10% Power Level (%): 95% Acceptable Drop out %: 10% N per Group: 42 (not taking into account drop out). N per Group: 47 (accounting for drop out). Total N: 141 subjects to be recruited.

4e. Sampling Technique: Randomized and open label. The investigators will randomly assign first patient into group A that is control group (warfarin group) then next patient to group B (rivaroxaban group) and then next patient into group C (Apixaban group). The investigators will repeat the cycle to achieve the target sample size in each group. Patients will be randomized in group A, B and C in a ratio of 1:1:1, to either control group A (Warfarin group with dose adjusted, target INR 2-3), group B (Rivaroxaban 20mg QD) and group C (Apixaban 5mg BD (bis in die i.e. Twice a day) or 2.5mg BD if having two or more of the following, patients with age ≥80years and/or creatinin≥1.5 and/or body weight ≤60kg). LVT resolution will be assessed by blinded cardiologist via transthoracic echocardiogram at 1, 3 and 6 months' interval after starting on the respective regimen.

5. DATA COLLECTION PROCEDURE: On a preformed proforma.

6. DATA ANALYSIS PROCEDURE: Stata version 14.2 will be used for data analysis. Frequencies with percentages will be reported for categorical variables. Means with standard deviation (depending on the normality assumption) or Median with Interquartile range (if the normality assumption is not met). The chi2-Square test will be used to assess the statistical significance for categorical variables (Fischer Exact test will be used if the expected cell count is >= 5). Independent Student t-test will be used to assess the statistical significance of continuous variables.

P-value ≤0.05 will be considered significant.

ELIGIBILITY:
Inclusion criteria

* All hemodynamically stable patients with LV thrombus on echocardiogram after.

Exclusion criteria

* Chronic Liver Disease (CLD) patients
* Creatinine clearance less than 15ml/min
* Recent Hemorrhagic stroke
* Thrombocytopenia, platelets <50k or anemia with baseline HB <9mg/dl
* Recent Major GI bleed
* History of atrial fibrillation and mitral stenosis
* History of deep vein thrombosis/pulmonary embolism and Patients already on anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Successful resolution of LV thrombus by Rivaroxaban and Apixaban in comparison to Warfarin | Within 6months of randamization
  Presence or absence of LV thrombus at one, three and six months follow up on echocardiogram.

SECONDARY OUTCOMES:
Time from start of drug to thrombus resolution in months | Within 6 months of randomization
  Secondary end point will be time in months after starting on drugs to LVT resolution (which will be assessed by follow up echocardiogram at one, three and six months duration)
No of events of major bleeding (defined by International Society of Thrombosis and Hemostasis criteria) | Within 6 months of randomization
  Number of events of major bleedings (defined by International Society of Thrombosis and Hemostasis criteria as, (a) a fall in hemoglobin level of 2 g/dL or more or documented transfusion of at least 2 units of packed red blood cells, (b) involvement of a critical anatomical site (intracranial, spinal, ocular, pericardial, articular, intramuscular with compartment syndrome, retroperitoneal) in all three groups of patients after starting on drugs till resolution of thrombus and/or maximum 6 months follow up after start of therapy if failed to resolve thrombus.
No of events of stroke (both ischemic and hemorrhagic) | Within 6 months of randomization
  No of events of stroke (both ischemic and hemorrhagic) in all three groups of patients after starting on drugs till resolution of thrombus and/or maximum 6 months follow up, after start of therapy if failed to resolve thrombus.

CONTACTS AND LOCATIONS:
Overall Officials: Ihsan Ullah, MD, Principal Investigator — Peshawar Institute of Cardiology
Locations (1):
- Peshawar Institute of Cardiology, Peshawar, KPK, Pakistan